CLINICAL TRIAL: NCT01714401
Title: The Development of Procedures to Optimalize the Intensive Care Units Patients Clinical Condition. Evaluation of Influence of Nebulized Bronchodilatory Drugs on Cardiac Repolarization
Brief Title: Nebulized Bronchodilators and Cardiac Repolarization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Radoslaw Owczuk, associate professor, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: TJ-1
Record Dates: First submitted 2012-10-23; First posted 2012-10-25 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Influence of Nebulized Bronchodilatators on Selected; Electrophysiological Parameters
MeSH Terms: interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Salbutamol 2,5 mg (Active Comparator): 25 mechanically ventilated patients to receive 2,5mg of nebulised salbtamol (Ventolin) duration of nebulisation - 20 minutes
  Interventions: Drug: Salbutamol 2,5 mg
- Salbutamol 5mg (Active Comparator): 25 mechanically ventilated patients 5 mg of nebulised salbutamol (Ventolin) duration of nebulisation - 20 minutes
  Interventions: Drug: Salbutamol 5mg

INTERVENTIONS:
Drug: Salbutamol 2,5 mg — 20 min nebulization of 2.5 mg of salbutamol
  Other Names: Ventolin 2.5mg
  Arms: Salbutamol 2,5 mg
Drug: Salbutamol 5mg — 20 min nebulization of 5 mg of salbutamol
  Other Names: Ventolin 5mg
  Arms: Salbutamol 5mg

SUMMARY:
Patients of the ICU's often require bronchodilatory treatment due to bronchospasm caused by conditions like : acute respiratory distress syndrome (ARDS), chronic obstructive pulmonary disease (COPD) or asthma. The β2 adrenergic drugs are one of the most commonly used for this purpose. However it is known that they may cause tachycardia and may have substantial proarrhythmic effect. The investigators' aim is to estimate the influence of nebulized bronchodilatory drugs on selected electrophysiological parameters, whose changes are generally recognized as potentially increasing the risk of ventricular and supraventricular arrhythmias. Two drugs will be compared - salbutamol given in two doses and ipratropium bromide

DETAILED DESCRIPTION:
50 mechanically ventilated patients above 18 years of age and with presence of clinical features of bronchospasm requiring treatment with nebulised short-acting beta-2 mimetic.

Participants will be randomly allocated into two equal groups: a group that was to receive the dose of 2.5 mg and a group that was to receive the dose of 5 mg of nebulised salbutamol. The duration of nebulisation will be set for 20 minutes and Holter ECG data are to be recorded for 60 minutes from the initiation of the nebuliser. The acquired Holter ECG data will be analysed at 10 time points: before salbutamol administration and 5, 10, 15, 20, 25, 30, 40, 50, and 60 minutes following initiation of nebulisation. Changes in QT interval, corrected QT intervals calculated using Bazett's correction and the Framingham formula and transmural dispersion of repolarization TDR will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* the necessity of b2 adrenergics an m2 mimetics administration

Exclusion Criteria:

* patients with past medical history of ventricular arrhythmias ( ventricular tachycardia, ventricular fibril, Torsade de pointes)
* patients with persistent atrial fibrillation
* patients with abnormal plasma sodium, potassium, magnesium, and ionized calcium concentration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2013-05-30 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
QT interval | one hour
  changes of QT interval after salbutamol nebulisation
corrected QT (QTc) interval using Bazett's (QTcB) correction | one hour
  changes of QTc interval after salbutamol nebulisation
corrected QT (QTc) interval using Framingham (QTcF) correction | one hour
  changes of QTc interval after salbutamol nebulisation
Tpeak-Tend | one hour
  changes in transmural dispersion of repolarization after salbutamol nebulisation

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Jasiński, MD, Principal Investigator — Medical University of Gdansk
Locations (2):
- Poland (2):
  - Medical University of Gdansk - Departament of Anesthesiolog and Intensive cCre, Gdansk
  - Medical University of Gdańsk - Departament of Anesthesiology and Intensive Care, Gdansk

REFERENCES:
- [Derived] Jasinski T, Owczuk R, Wujtewicz M. The effect of nebulized salbutamol on atrial electrical properties in mechanically ventilated critically ill patients - a randomized, double-blind study. Anaesthesiol Intensive Ther. 2018;50(4):270-276. doi: 10.5603/AIT.a2018.0031. Epub 2018 Sep 22. PMID 30242825